CLINICAL TRIAL: NCT04543578
Title: Evaluation of the Applicability and Effectiveness of a Protocol for the Multidisciplinary Management of Acute Cholecystitis
Brief Title: Evaluation of a Protocol for Multidisciplinary Management of Acute Cholecystitis.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundacion Miguel Servet (Other)
Responsible Party: Sponsor
Other Study IDs: DIGESTIVO CHN-VBP
Record Dates: First submitted 2020-09-02; First posted 2020-09-10 (Actual); Last update posted 2020-12-14 (Actual); Status verified 2020-12

CONDITIONS: Acute Cholecystitis
Keywords: Acute cholecystitis; EUS-guided cholecystostomy; Percutaneous cholecystostomy; Laparoscopic cholecystectomy
MeSH Terms: conditions — Cholecystitis, Acute

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Patients unfit for Surgery with mild-moderate acute cholecyst: Conservative treatment (antibiotics, etc). EUS-guided gallbladder drainage will be considered in recurrent acute cholecystitis and in patients with no improvement in 48-72h after admission.
- Patients unfit for Surgery with severe acute cholecystitis: Percutaneous cholecystostomy or Endoscopic Ultrasound (EUS)-guided cholecystostomy (the latter is not 24/7 available). Palliative care may also be considered in patients with very serious conditions and low life expectancy.
- Patients suitable for Surgery with high and intermediate risk: Admission in Gastroenterology Department. antibiotic treatment. Close follow-up of posible AC complications. Once choledocholithiasis is solved or ruled our, the patient will be considered for same-admission cholecystectomy or programmed cholecystectomy.
  * High risk: Endoscopic Retrograde Cholangiopancreatography (ERCP) will be performed.
  * Intermediate risk: EUS or Magnetic Resonance Cholangiopancreatography prior to consider ERCP.
- Patients suitable for Surgery with low risk: Admission in Surgery Department. According to the AC severity:
  * Mild-moderate AC: check de ASA/Charlson comorbidity index.
  * ASA I-II/Charlson <6: laparoscopic cholecystectomy
  * ASA > =III/Charlson >=6: close follow-up 24-48h. Consider laparoscopic cholecystostomy (if no improvement is achieved)
  * Severe AC: consider Intensive Care Unit admission. Percutaneous cholecystectomy.

SUMMARY:
Acute cholecystitis is a complex disease and its management is sometimes controversial. Two main factors contribute to its complexity: the patient's surgical risk and the possibility of concomitant choledocholithiasis. The design of a multidisciplinary protocol between the services of Gastroenterology and Surgery aims to harmonize its management and to adapt it to the most recent guidelines. As it concerns more than one department, it is crucial to analyze its compliance and effectiveness.

DETAILED DESCRIPTION:
Adult patients attending the emergency department and diagnosed with acute cholecystitis will be asked to participate. Those considered not suitable for surgery will be admitted in a medical department and assigned to conservative treatment or cholecystostomy, according to their acute cholecystitis severity. In patients suitable for surgery, risk of concomitant choledocholithiasis will be assessed and patients will be assigned to low risk or intermediate-high risk. The latter will be admitted in a medical department, and choledocholithiasis will be ruled out and treated if present. The former will be offered cholecystectomy or cholecystostomy according to their surgical risk and acute cholecystitis severity. A flowchart with extended information is attached.

PRIMARY OBJECTIVES

• To harmonize the management of acute cholecystitis with a multidisciplinary protocol based on the most recent guidelines.

SECONDARY OBJECTIVES

* To analyze the compliance with this protocol.
* To evaluate the validity of the criteria used in the decision-making process.
* To assess the morbidity and mortality of different groups of patients according to the selected treatment, severity of cholecystitis and baseline characteristics of the patient.
* To estimate the resource use in each group of patients.
* To compare current data with a previous period.
* To adapt and modify the protocol according the study results. INCLUSION CRITERIA
* Patients aged 18 or older who agree to participate (an informed consent signature is required)
* Patients attended in the emergency department of our hospital and diagnosed with acute cholecystitis according to the Tokyo criteria.

EXCLUSION CRITERIA

* Patients under 18 years or patients who refuse to participate in the study
* Patients diagnosed with acute cholangitis during admission for other causes.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 or older who agree to participate (an informed consent signature is required)
* Patients attended in the emergency department of our hospital and diagnosed with acute cholecystitis according to the Tokyo criteria.

Exclusion Criteria:

* Patients under 18 years or patients who refuse to participate in the study
* Patients diagnosed with acute cholangitis during admission for other causes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients attended in the emergency department of CHN and diagnosed with acute cholecystitis.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-07 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Inclusion rate | During inclusion period
  Rate of patients with AC diagnosis registered in the study
Protocol compliance | During inclusion period
  Rate of patients with complete protocol compliance
Morbidity in the different subtypes of patients | three months after hospital discharge
  length of hospital stay, need for unplanned readmissions, recurrent cholecystitis
Mortality in the different subtypes of patients | three months after hospital discharge
  90-day disease-specific mortality

SECONDARY OUTCOMES:
Protocol compliance failure | every 3 months throughout study completion (up to 1 year)
  Identify causes of protocol compliance failure
Evaluate the technical success | During inclusion period (up to 1 year)
  Evaluate clinical success and adverse events of the different treatments.
Evaluate the accuracy in the diagnosis | three months after hospital discharge or after ERCP
  Evaluate the accuracy of Magnetic Resonance Cholangiopancreatography (MRCP) and EUS in the diagnosis of concomitant choledocholithiasis

CONTACTS AND LOCATIONS:
Overall Officials: Federico Bolado Concejo, MD, PhD, Principal Investigator — Complejo Hospitalario de Navarra
Locations (1):
- Complejo Hospitalario de Navarra, Pamplona, Navarre, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Yokoe M, Hata J, Takada T, Strasberg SM, Asbun HJ, Wakabayashi G, Kozaka K, Endo I, Deziel DJ, Miura F, Okamoto K, Hwang TL, Huang WS, Ker CG, Chen MF, Han HS, Yoon YS, Choi IS, Yoon DS, Noguchi Y, Shikata S, Ukai T, Higuchi R, Gabata T, Mori Y, Iwashita Y, Hibi T, Jagannath P, Jonas E, Liau KH, Dervenis C, Gouma DJ, Cherqui D, Belli G, Garden OJ, Gimenez ME, de Santibanes E, Suzuki K, Umezawa A, Supe AN, Pitt HA, Singh H, Chan ACW, Lau WY, Teoh AYB, Honda G, Sugioka A, Asai K, Gomi H, Itoi T, Kiriyama S, Yoshida M, Mayumi T, Matsumura N, Tokumura H, Kitano S, Hirata K, Inui K, Sumiyama Y, Yamamoto M. Tokyo Guidelines 2018: diagnostic criteria and severity grading of acute cholecystitis (with videos). J Hepatobiliary Pancreat Sci. 2018 Jan;25(1):41-54. doi: 10.1002/jhbp.515. Epub 2018 Jan 9. PMID 29032636
- [Background] Ansaloni L, Pisano M, Coccolini F, Peitzmann AB, Fingerhut A, Catena F, Agresta F, Allegri A, Bailey I, Balogh ZJ, Bendinelli C, Biffl W, Bonavina L, Borzellino G, Brunetti F, Burlew CC, Camapanelli G, Campanile FC, Ceresoli M, Chiara O, Civil I, Coimbra R, De Moya M, Di Saverio S, Fraga GP, Gupta S, Kashuk J, Kelly MD, Koka V, Jeekel H, Latifi R, Leppaniemi A, Maier RV, Marzi I, Moore F, Piazzalunga D, Sakakushev B, Sartelli M, Scalea T, Stahel PF, Taviloglu K, Tugnoli G, Uraneus S, Velmahos GC, Wani I, Weber DG, Viale P, Sugrue M, Ivatury R, Kluger Y, Gurusamy KS, Moore EE. 2016 WSES guidelines on acute calculous cholecystitis. World J Emerg Surg. 2016 Jun 14;11:25. doi: 10.1186/s13017-016-0082-5. eCollection 2016. PMID 27307785
- [Background] Chisholm PR, Patel AH, Law RJ, Schulman AR, Bedi AO, Kwon RS, Wamsteker EJ, Anderson MA, Elta GH, Govani SM, Prabhu A. Preoperative predictors of choledocholithiasis in patients presenting with acute calculous cholecystitis. Gastrointest Endosc. 2019 May;89(5):977-983.e2. doi: 10.1016/j.gie.2018.11.017. Epub 2018 Nov 19. PMID 30465770
- [Background] ASGE Standards of Practice Committee; Maple JT, Ben-Menachem T, Anderson MA, Appalaneni V, Banerjee S, Cash BD, Fisher L, Harrison ME, Fanelli RD, Fukami N, Ikenberry SO, Jain R, Khan K, Krinsky ML, Strohmeyer L, Dominitz JA. The role of endoscopy in the evaluation of suspected choledocholithiasis. Gastrointest Endosc. 2010 Jan;71(1):1-9. doi: 10.1016/j.gie.2009.09.041. No abstract available. PMID 20105473
- [Background] ASGE Standards of Practice Committee; Buxbaum JL, Abbas Fehmi SM, Sultan S, Fishman DS, Qumseya BJ, Cortessis VK, Schilperoort H, Kysh L, Matsuoka L, Yachimski P, Agrawal D, Gurudu SR, Jamil LH, Jue TL, Khashab MA, Law JK, Lee JK, Naveed M, Sawhney MS, Thosani N, Yang J, Wani SB. ASGE guideline on the role of endoscopy in the evaluation and management of choledocholithiasis. Gastrointest Endosc. 2019 Jun;89(6):1075-1105.e15. doi: 10.1016/j.gie.2018.10.001. Epub 2019 Apr 9. PMID 30979521
- [Background] Manes G, Paspatis G, Aabakken L, Anderloni A, Arvanitakis M, Ah-Soune P, Barthet M, Domagk D, Dumonceau JM, Gigot JF, Hritz I, Karamanolis G, Laghi A, Mariani A, Paraskeva K, Pohl J, Ponchon T, Swahn F, Ter Steege RWF, Tringali A, Vezakis A, Williams EJ, van Hooft JE. Endoscopic management of common bile duct stones: European Society of Gastrointestinal Endoscopy (ESGE) guideline. Endoscopy. 2019 May;51(5):472-491. doi: 10.1055/a-0862-0346. Epub 2019 Apr 3. PMID 30943551
- [Background] Luk SW, Irani S, Krishnamoorthi R, Wong Lau JY, Wai Ng EK, Teoh AY. Endoscopic ultrasound-guided gallbladder drainage versus percutaneous cholecystostomy for high risk surgical patients with acute cholecystitis: a systematic review and meta-analysis. Endoscopy. 2019 Aug;51(8):722-732. doi: 10.1055/a-0929-6603. Epub 2019 Jun 25. PMID 31238375

DOCUMENTS (1):
  • Study Protocol (2020-09-28): https://cdn.clinicaltrials.gov/large-docs/78/NCT04543578/Prot_000.pdf